CLINICAL TRIAL: NCT06699693
Title: Effectiveness of Ultrasonography-guided Pericapsular Nerve Group Block in Patients With Adhesive Capsulitis Resistant to Conservative Treatment
Brief Title: Effectiveness of Ultrasonography-guided Pericapsular Nerve Group Block in Patients With Adhesive Capsulitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Bora Uzuner, Assistant Professor, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (No:223/2024)
Record Dates: First submitted 2024-11-17; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Pericapsular Nerve Group Block (PENG Block); Kinesiophobia; Adhesive Capsulitis and Frozen Shoulder Syndrome
Keywords: Adhesive capsulitis; Pericapsular Nerve Group Block; pain; function; kinesiophobia
MeSH Terms: conditions — Kinesiophobia; Bursitis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 Injection+Mobilization (Active Comparator): Group 1 patients underwent ultrasound-guided PENG block (20 cc of a solution containing 0.25% bupivacaine hydrochloride and 6 mg betamethasone) by an experienced algologist (BU) before starting mobilization treatment
  Interventions: Procedure: ultrasonography-guided PENG block
- Group 2 Mobilization (Active Comparator): only mobilization therapy on shoulder pain, function, and kinesiophobia in patients with AC resistant to conservative treatment,
  Interventions: Other: Mobilization

INTERVENTIONS:
Procedure: ultrasonography-guided PENG block — This study aimed to evaluate the effect of ultrasonography-guided PENG block prior to joint mobilization therapy on shoulder pain, function, and kinesiophobia in patients with AC resistant to conservative treatment, in comparison with a control group
  Arms: Group1 Injection+Mobilization
Other: Mobilization — The mobilization methods encompassed the scapula and clavicular joints, in addition to the glenohumeral (GH) joint, taking into consideration their biomechanical interactions. These exercises were supervised and administered by the physiotherapist during each session. Additionally, the patients were provided with a home exercise program that included exercises for posture, thera band, and finger ladder, with instructions to perform 10-15 repetitions twice a day independently [
  Arms: Group 2 Mobilization

SUMMARY:
We aimed to observe the effects of Ultrasound-Guided Pericapsular Nerve Group Block administered before joint mobilization therapy on shoulder pain levels, function, and kinesiophobia in patients with resistant Adhesive Capsulitis.

Voluntary patients who applied to the Physical Therapy and Algology Department, did not benefit from physical therapy, and were recommended injection and mobilization therapy will be included in the study. Patients who decline injection but consent to mobilization therapy will be included as the control group. Those who accept the injection will be treated as Group 1 (Block + mobilization therapy), and those who decline the injection will be treated as Group 2 (mobilization therapy only).

Group 1 patients will receive a pericapsular nerve block before mobilization therapy, and a one-hour observation period will follow to assess the effectiveness of the procedure and monitor the patient. Patients will be evaluated for pain and range of motion (ROM) before and after the injection. Subsequently, they will undergo mobilization therapy three times a week for six weeks. Group 2 will follow the same program but will only receive mobilization therapy.

The following demographic data will be collected from the patients included in the study: age, gender, height, weight, education level, occupation, employment status, history of alcohol and smoking, comorbidities, current medications, dominant hand, and exercise status.

Patients' medical histories will be reviewed, and any prior test results (e.g., blood glucose, thyroid dysfunction, lipid levels, vitamin D, and vitamin B12 levels) will be recorded. Findings from previous diagnostic or differential diagnostic imaging for shoulder pain (shoulder X-rays, ultrasound, or MRI) as well as routine biochemistry blood test results will be evaluated and documented. Comprehensive physical examinations, including systemic and neurological assessments, ROM measurements, and muscle strength evaluations, will also be conducted.

* **DASH Score (Disabilities of the Arm, Shoulder, and Hand Questionnaire):** This questionnaire consists of three sections. Among the 30 questions, 21 assess difficulty in daily living activities, 5 address pain, activity-related pain, tingling, stiffness, and weakness, while 4 evaluate social function, work, sleep, and self-confidence. All questions are rated on a 5-point Likert scale, where 5 indicates extreme difficulty. Higher scores reflect greater disability.
* **Modified Constant-Murley Score:** This score evaluates four parameters with a total of 100 points. Pain is allocated 15 points, daily living activities 20 points, muscle strength 25 points, and shoulder ROM (elevation, external rotation, abduction, internal rotation) 40 points. Higher scores indicate better function.
* **VAS (Visual Analog Scale) for Pain:** Pain is scored as rest VAS, movement-related VAS, and night pain VAS on a scale from 0 to 10, where 0 indicates no pain and 10 indicates the highest level of pain.
* **Tampa Scale of Kinesiophobia:** A 17-item scale developed to measure fear of movement and re-injury. It includes parameters such as work-related activities, fear of injury/re-injury, and fear-avoidance behavior.
* **Shoulder Range of Motion (ROM):** Measured in degrees using a goniometer and recorded.
* **Complications and Side Effects:** These will be inquired from the patient and recorded.

  * **Ultrasound-Guided Pericapsular Nerve Group Block:** This procedure will be performed in an outpatient clinic setting and applied only once to Group 1.

During the procedure, with the patient's arm in an externally rotated and 45-degree abducted position, a linear ultrasound probe will be placed longitudinally between the coracoid process and the humeral head. After identifying the humeral head, the subscapularis muscle tendon and the overlying deltoid muscle will be visualized. A 50 mm needle will be advanced using an in-plane technique into the area between the deltoid muscle and subscapularis tendon. A total of 20 cc of a solution containing 0.25% bupivacaine hydrochloride and 6 mg of betamethasone (Celestone Chronodose) will be injected.

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder pain (Visual Analog Scale, VAS: 50 mm or more) and limitation of movement (at least 50% loss in active and passive ROM on the affected side) for at least 3 months
2. Poor response to previous exercise and drug therapy

Exclusion Criteria:

1. Severe systemic illnesses such as neurological diseases (e.g., Parkinson's disease, previous cerebrovascular disease, dementia), psychiatric disorders (e.g., major depression), diabetes mellitus, malignancy, infection, rheumatologic diseases (e.g., systemic lupus erythematosus), neuromuscular diseases (e.g., motor neuron diseases)
2. History of major orthopedic surgery, such as total shoulder replacement
3. History of steroid injection into the shoulder within the last 3 months
4. Previous mobilization therapy on the affected shoulder
5. Advanced-stage heart, liver, or kidney failure
6. High risk of bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Pain | for 6 weeks
  Resting pain, pain during activity, and night pain were assessed using VAS, where 0 indicated no pain and 10 represented the highest pain level
Shoulder Joint Range of Motion (ROM) | for 6 weeks
  Active and passive shoulder flexion, abduction, internal rotation, and external rotation were measured with the patient lying supine, using a goniometer
Function | for 6 weeks
  Disabilities of Arm, Shoulder and Hand (DASH)
  This questionnaire consists of 3 parts. Twenty-one of the 30 questions are about difficulty in activities of daily living, 5 questions are about pain, activity-related pain, tingling, stiffness and weakness, and 4 questions are about social function, work, sleep and self-confidence. All questions are rated on a Likert scale of 5, where 5 indicate too much difficulty. A high score indicates limitation. Turkish validity and reliability were examined
Function | for 6 weeks
  Modified Constant-Murley Score (MCMS) The four parameters are evaluated with a total of 100 points. Pain is calculated as 15 points, activities of daily living 20 points, muscle strength 25 points, and shoulder ROM (elevation, ER, Abd, IR) 40 points and high scores indicate good function. Turkish validity and reliability were investigated
Muscle strength | for 6 weeks
  Muscle strength was measured using a portable hand dynamometer
Kinesiophobia | for 6 weeks
  The Tampa Scale of Kinesiophobia (TSK): The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia. The Turkish version was validated and is reliable

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty, Ondokuz Mayis University, Samsun, Turkey, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263